CLINICAL TRIAL: NCT05944198
Title: Clinical Study of 18F-labeled Probes Targeting Fibroblast Activating Protein and Integrin avβ3 (FAPI-RGD) to Assess Disease Activity in Rheumatoid Arthritis
Brief Title: Clinical Study of 18F-FAPI-RGD PET/CT in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Wang, Associate senior physician, Sichuan Provincial People's Hospital
Other Study IDs: SichuanPPH-RA
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about 18F-FAPI-RGD PET/CT imaging in assessing rheumatoid arthritis disease activity. Participants will undergo clinical evaluation and 18F-FAPI-RGD PET/CT examination.

DETAILED DESCRIPTION:
Patients with rheumatoid arthritis who met the 2010 American College of Rheumatology/European League against Rheumatism Rheumatoid arthritis classification criteria will be included. All patients will be assessed for disease activity and the clinical disease activity Index (cDAI) was calculated. Blood sedimentation rate and CRP assay results will be collected. All patients will undergo 18F-FAPI-RGD PET/CT examination. The correlation of cDAI, ESR and CRP levels with PET joint count and PET joint index as measured by 18F-FAPI-RGD PET/CT will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis who meet the 2010 American College of Rheumatology/European League Against Rheumatism Rheumatoid arthritis classification criteria.

Exclusion Criteria:

* A. Patients with malignant tumors and other rheumatic immune diseases; B. clinical and conventional radiographic inspection of materials; C. researchers think not suitable for other information to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rheumatoid arthritis who meet the 2010 American College of Rheumatology/European League Against Rheumatism Rheumatoid arthritis classification criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Correlation between clinical indicators and PET/CT results | 1 month
  Correlation of clinical disease activity Index (cDAI), erythrocyte sedimentation rate (ESR), and CRP levels with 18F-FAPI-RGD PET/CT results

CONTACTS AND LOCATIONS:
Locations (1):
- Departments of Nuclear Medicine, Sichuan Provincial People's Hospital, Chengdu, Sichuan, China